CLINICAL TRIAL: NCT01551992
Title: Affixing Polypropylene Mesh Using Barbed Suture (Quill™ Srs) During Laparoscopic Sacrocolpopexy Randomized Controlled Trial
Brief Title: Affixing Polypropylene Mesh Using Barbed Suture (Quill™ Srs) During Laparoscopic Sacrocolpopexy Randomized Controlled Trial (Quill Lsc)
Acronym: QUILL-LSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Quill LSC
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Prolapse
Keywords: Sutures; Pelvic Organ Prolapse; Sacrocolpopexy; Laparoscopy
MeSH Terms: conditions — Prolapse; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interrupted suture (Active Comparator): interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA)
  Interventions: Procedure: Quill suture vs. Interrupted suture
- Quill suture (Active Comparator): self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada)
  Interventions: Procedure: Quill suture vs. Interrupted suture

INTERVENTIONS:
Procedure: Quill suture vs. Interrupted suture — To compare two methods of polypropylene mesh attachment during laparoscopic sacrocolpopexy (LSC): running technique using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

SUMMARY:
1.0 STUDY OBJECTIVE 1.1 PRIMARY OBJECTIVE - To compare two methods of polypropylene mesh attachment during laparoscopic sacrocolpopexy (LSC): running technique using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

1.2 SECONDARY OBJECTIVE - To compare laparoscopic sacrocolpopexy anatomic failure rates at 6 months post-operative follow-up using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA). The investigators will also assess mesh erosion rates, costs, and surgeon satisfaction rates.

2.0 HYPOTHESIS 2.1 Primary: 2.1.a. Attachment of mesh using the running technique with self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) will be faster than the standard fixation interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

2.2 Secondary: 2.2.a. Attachment of mesh using the running technique with self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) will be less costly than the standard fixation interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA).

2.2.b. Failure rates and mesh erosion rates for each technique will be equally low.

2.2.c. Surgeons will prefer the barbed running technique over the interrupted technique based on subjective surgeon satisfaction questionnaires.

ELIGIBILITY:
INCLUSION CRITERIA

* >18 years old
* Undergoing LSC with or without other procedures for pelvic organ prolapse or incontinence
* Willing to return for follow-up visits
* Written informed consent obtained from each subject
* Must be having a robotic assisted laparoscopic sacrocolpopexy

Exclusion Criteria:

* Decline to participate
* Pregnant or contemplating future pregnancy
* Unable to participate in the informed consent process

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Mesh attachment interval | Intraoperatively
  To compare two methods of polypropylene mesh attachment during laparoscopic sacrocolpopexy (LSC): running technique using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus interrupted technique using 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA)in terms of time.

SECONDARY OUTCOMES:
Anatomic outcomes using the two suture types | 6 months post-operatively
  To compare laparoscopic sacrocolpopexy anatomic failure rates at 6 months post-operative follow-up using self-anchoring 1 barbed delayed absorbable suture (Quill™ SRS, Angiotech Pharmaceuticals, Inc. Vancouver, Canada) versus 0 non-barbed delayed absorbable suture (PDS II™, Ethicon, Somerville, NJ, USA). We will also assess mesh erosion rates, costs, and surgeon satisfaction rates.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente San Diego, San Diego, California, United States

REFERENCES:
- [Derived] Tan-Kim J, Nager CW, Grimes CL, Luber KM, Lukacz ES, Brown HW, Ferrante KL, Dyer KY, Kirby AC, Menefee SA. A randomized trial of vaginal mesh attachment techniques for minimally invasive sacrocolpopexy. Int Urogynecol J. 2015 May;26(5):649-56. doi: 10.1007/s00192-014-2566-8. Epub 2014 Nov 25. PMID 25421934